CLINICAL TRIAL: NCT05584709
Title: A Phase 1B, Open-Label, Dose-Escalation Study of the Safety and Efficacy of an Anti-CD38 Antibody Drug Conjugate (STI-6129) in Patients With Advanced Solid Tumors
Brief Title: Study to Access Anti-CD38 Anibody Drug in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 38ADC-AST-101
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-6129 infusion (Experimental): Intravenous infusion to be given with prophylaxis for infusion reactions if necessary.
  Interventions: Biological: STI-6129

INTERVENTIONS:
Biological: STI-6129 — Repeated 4-week intravenous infusion cycles of STI-6129 will be given. (one infusion every four weeks).
  Other Names: Anti-CD38 antibody drug conjugate

SUMMARY:
This study is a Phase 1b, single-center, open-label, dose-finding trial designed to identify the Recommended Phase 2 Dose (RP2D) of STI 6129 by assessing the safety, preliminary efficacy, and immunogenicity in subjects with any advanced solid tumor.

The patients that will be treated with STI-6129 in this trial are advanced solid tumor patients who have received prior lines of treatment.

DETAILED DESCRIPTION:
The study is a sequential cohort ascending dose (3+3 methodology after a sentinel at the 0,25 mg/kg level) study to confirm safety and identify DLTs in the study population and determine the maximum tolerated dose (MTD) and the RP2D.

The range of proposed doses includes optimal doses identified in parallel safety studies of STI-6129 for the treatment of relapsed/refractory systemic amyloid light chain (AL) amyloidosis that are currently ongoing (a three-stage, multicenter, open-label, dose -finding, Phase 1 trial to identify the RP2D). STI-6129 will be given as an intravenous (IV) infusion.

Each patient enrolled will received repeated 4-week cycles of STI-6129 (Q4W) Total duration will vary according to patient response. After the treatment period, patients will be monitored for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumors, such as but not limited to:

  * Lung squamous cell carcinoma (LSCC)
  * Esophageal squamous cell carcinoma (ESCC)
  * Head and neck squamous cell carcinoma (HNSCC)
  * Microsatellite stable colorectal cancer (MSS-CRC) that are refractory to standard therapy (to include standard chemotherapy and anti-PD-L1 therapy concurrently or sequentially prior to enrollment) or for which standard or curative therapy does not exist or is not considered appropriate by the Investigator. Patients with MSS-CRC must have completed at least 2 lines of standard of care treatments prior to enrollment.
* Adequate hematologic (with no blood product or hematopoietic growth factor support during the prior 7 days), renal and hepatic function, as defined by the following laboratory values; test performed within 7 days prior to first dose of STI-6129:

  a. Hematologic: i. Absolute neutrophil count (ANC) ≥ 1000 cells/μL ii. Platelet count ≥ 50,000 platelets/μL iii. Hemoglobin (Hgb) ≥ 8.0 g/dL b. Renal: creatine clearance (CrCl) ≥ 60 mL/min by Cockroft-Gault formula (Protocol Appendix 1) c. Hepatic: i. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ˂ 3x the upper limit of normal (ULN) ii. serum total bilirubin ˂ 1.5x ULN (except for patients in whom hyperbilirubinemia is attributed to Gilbert's Syndrome) iii. Alkaline phosphatase times ˂ 3x ULN (˂ 5 times ULN if considered due to tumor)
* ECOG performance status of 0 or 1
* Be willing and able to comply with the study schedule and all other protocol requirements
* Willing to follow contraception guidelines

Exclusion Criteria:

* Use of systemic anti-tumor therapy or an investigational drug within 5 half-lives or 4 weeks of D1 whichever is shorter, preceding the first dose of study drug.
* Received any prior anti-CD38 treatment within 90 days.
* A diagnosis of other malignancies that have required systemic therapy within the last 3 years or is not in complete remission. Exceptions are non-metastatic basal cell or squamous cell carcinomas of the skin or prostate cancer or in situ cancer that does not require treatment or is well under control.
* A current history of CTCAE Grade 3 muscle paresis, eyelid conditions, glaucoma controlled with medication or watering eyes or any other ocular disorder that is CTCAE Grade 2.
* A history of a dose-limiting immune-related adverse event during PD-1 axis blockade.
* INR or aPTT > 1.5 times ULN within one week prior to the infusion of STI-6129, unless on a stable dose of an anticoagulant
* Patients with ≥ Grade 3 neuropathy or Grade 2 neuropathy with associated pain.
* New York Heart Association (NYHA) Class > 2.
* QTcF > 470 msec on a 12-lead ECG.
* Treatment with potent inhibitors of cytochrome P450 systems: CYP3A4, CYP2B6 and CYP1A2, or strong inhibitors or transducers of transporter P-glycoprotein (Pgp or MDR1) or breast cancer resistance protein (BCRP or ABCG2) during the study. See https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers for details.
* Symptomatic, untreated brain metastases. Patients with treated brain metastases may be treated at least 1 week after gamma knife stereotactic radiation or at least 2 weeks after whole brain radiation if symptoms have recovered with discontinuation of steroids. Patients with small, asymptomatic brain metastases may be considered for enrollment.
* Symptomatic CNS disease (i.e. cord compression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events by type, frequency, severity, and causality (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of adverse events (AEs) by type, frequency, severity, and causality
Incidence of serious adverse events by type, frequency, severity, and causality (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of serious AEs (SAEs) by type, frequency, severity, and causality
Incidence of dose-limiting toxicities (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of dose-limiting toxicities
Incidence of neurotoxicity (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of neurotoxicity
Incidence of laboratory abnormalities (safety) | Baseline through study completion at up to approximately 24 months
  Safety as assessed by incidence of laboratory abnormalities using the Common Terminology Criteria for Adverse Events (CTCAE Version 5)

SECONDARY OUTCOMES:
Evaluation of response rate | Baseline through study completion at up to approximately 24 months
  Evaluation of response rate for advanced solid tumors using Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
Overall response | Baseline through study completion at up to approximately 24 months
  Response assessed according to the Evaluation Criteria in Solid Tumors (RECIST v1.1)
Overall duration | Baseline through study completion at up to approximately 24 months
  Duration assessed according to the Evaluation Criteria in Solid Tumors (RECIST v1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States